CLINICAL TRIAL: NCT01817556
Title: A Multicenter, Active-controlled, Randomized, Double-blind Paralleled-group Clinical Trial to Evaluate the Efficacy of 4-week Treatment With Stillen Tab. in Patients With Acute or Chronic Gastritis
Brief Title: A Study to Evaluate the Efficacy and of Stillen Tab. and to Demonstrate the Non-inferiority of Stillen Tab.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA9601_Gas_IV
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Acute Gastritis; Chronic Gastritis
MeSH Terms: interventions — DA 9601

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stillen Tab. (Experimental): administered three times daily for four weeks
  Interventions: Drug: Stillen Tab.
- Mucosta Tab. (Active Comparator): administered three times daily for four weeks
  Interventions: Drug: Mucosta Tab.

INTERVENTIONS:
Drug: Stillen Tab.
  Arms: Stillen Tab.
Drug: Mucosta Tab.
  Arms: Mucosta Tab.

SUMMARY:
This is a multicenter, active-controlled, randomized, double-blinded, paralleled group clinical study to evaluate the efficacy of 4-week treatment with Stillen tab. in patients with acute or chronic gastritis. Subject will receive Stillen tab or Mucosta tab., three times a day for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age is over 20 years old, under 75 years old, men or women
* Patients diagnosed with acute or chronic gastritis by gastroscopy
* Patients with one or more erosions found by gastroscopy
* Signed the informed consent forms

Exclusion Criteria:

* Patients with peptic ulcer and gastroesophageal reflux disease
* Patients administered with prokinetics, H2 receptor antagonists, proton pump inhibitors, anticholinergic drugs or non-steroid anti-inflammatory drugs prior to study in 2 weeks
* Patients with surgery related to gastroesophageal
* Patients with Zollinger-Ellison syndrome
* Patients with any kind of malignant tumor
* Patients administered with anti-thrombotic drugs
* Patients with significant cardiovascular, pulmonary, heptic, renal, hemopoietic or endocrine system primary disease
* Women either pregnant or breast feeding

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Improvement rates of erosive gastritis | 4 weeks
  Improvement rates of erosive gastritis (%)
  = (improved cases)/(total cases administered) * 100

SECONDARY OUTCOMES:
Healing rates of erosive gastritis | 4 weeks
  Healing rates of erosive gastritis (%)
  = (healed cases)/(total cases administered)*100
Symptoms improved level | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chan Lee, M.D., Ph.D., Principal Investigator — Yonsei University, Severance Hospital of Korea; Jin Il Kim, M.D., Ph.D., Principal Investigator — The Catholic University, Yeouido St. Mary's Hospital of Korea; Kwang Ro Joo, M.D., Ph.D., Principal Investigator — Kyung Hee University Gangdong Hospital of Korea; Dong Il Park, M.D., Ph.D., Principal Investigator — Kangbuk Samsung Hospital of Korea; In Kyung Sung, M.D.,Ph.D., Principal Investigator — Konkuk University Hospital of Korea; Kyu Chan Huh, M.D., Ph.D., Principal Investigator — Konyang University Hospital of Korea; Jung Il Suh, M.D., Ph.D., Principal Investigator — Dongguk University Gyeongju Hospital of Korea; Su Jin Hong, M.D., Ph.D., Principal Investigator — Soon Chun Hyang University Bucheon Hospital of Korea; Jin Heung Kim, M.D., Ph.D., Principal Investigator — Ajou University Hospital of Korea; Dae Hwan Kang, M.D., Ph.D., Principal Investigator — Pusan National University Yangsan Hospital of Korea; Tae Joo Jeon, M.D., Ph.D., Principal Investigator — Inje University Sanggye Paik Hospital of Korea; Tea Oh Kim, M.D., Ph.D., Principal Investigator — Inje University Haeundae Paik Hospital of Korea; Hyun Yong Jeong, M.D., Ph.D., Principal Investigator — Chungnam National Unviersity Hospital of Korea
Locations (1):
- Yonsei University Health System, Severance Hospital, IRB, Seoul, South Korea